CLINICAL TRIAL: NCT02108847
Title: Ultrasound Guided Fascia Iliaca Block for Postoperative Analgesia After Elective Total Hip Arthroplasty
Brief Title: Ultrasound Guided Fascia Iliaca Block for Pain Control After Elective Hip Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatoon Health Region (Other)
Responsible Party: Principal Investigator, Jacelyn Larson, M.D., University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Bio 13-314
Record Dates: First submitted 2014-03-21; First posted 2014-04-09 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Arthroplasty, Replacement, Hip; Fascia Iliaca Block
Keywords: Arthroplasty, Replacement, Hip; Pain, Postoperative; Nerve Block; Anesthesia, Regional; Fascia Iliaca Block; Ultrasound Guided
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fascia Iliaca Block - Ropivacaine (Experimental): Ultrasound guided fascia iliaca block performed preoperatively with 40 mL of 0.2% ropivacaine.
  Interventions: Drug: .2% Ropivacaine; Procedure: Fascia Iliaca Block
- Fascia Iliaca Block - Saline (Sham Comparator): Ultrasound guided fascia iliaca block performed preoperatively with 40 mL of Saline.
  Interventions: Drug: Saline; Procedure: Fascia Iliaca Block

INTERVENTIONS:
Drug: .2% Ropivacaine
  Arms: Fascia Iliaca Block - Ropivacaine
Drug: Saline
  Arms: Fascia Iliaca Block - Saline
Procedure: Fascia Iliaca Block — Ultrasound-guided regional anesthesia block to the groin area.

SUMMARY:
The purpose of this study is to determine whether ultrasound guided fascia iliaca blocks performed before surgery help to reduce pain after elective total hip replacements.

DETAILED DESCRIPTION:
Total hip arthroplasty is associated with moderate to severe pain in the acute postoperative period, which can increase the risk of postoperative complications such as thromboembolism, myocardial ischemia/infarction, pneumonia, poor wound healing, insomnia, and delirium.

Sensory innervation of the hip joint comes from a combination of peripheral nerves, including femoral, obturator, sciatic, superior gluteal, and nerve for the quadratus femoris muscle. Superficial innervation of the skin involved in incision for hip arthroplasty comes from the lateral femoral cutaneous nerve (LFCN).

The fascia iliaca block (FIB) was originally described in 1989 using a landmark technique. The ultrasound guided FIB was introduced in recent years, and has been shown to produce a better quality of block than the landmark technique. It appears to consistently block the femoral and LFCN, while being less successful in achieving consistent obturator blockade.

The FIB is effective for analgesia for hip fracture injuries in the emergency department. Thus far, there has been limited exploration into the potential use of this block as a tool for postoperative analgesia after elective hip arthroplasty. The potential benefits of this regional block, as with other regional techniques, include better analgesia, less opioid use and associated side effects, and an improved overall patient satisfaction with postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists' (ASA) score I, II or III
* Scheduled for elective total hip arthroplasty

Exclusion Criteria:

* Contraindication to regional anesthesia (allergy to local anesthetic, coagulopathy, infection or malignancy in the area)
* Neurologic disorder affecting the ability to sense pain
* Long term opioid use or chronic pain disorder
* History of drug or alcohol abuse
* Patient refusal
* Pregnancy
* Revision procedures
* General anesthetic
* Psychiatric or mental conditions that may affect assessment of outcomes

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Cumulative opioid consumption | 12 hours after surgery
  Dilaudid will be used for analgesia postoperatively. If there is a contraindication to Dilaudid, another opioid will be ordered for analgesia, and doses will subsequently be converted back to Dilaudid equivalent doses for comparison
Cumulative opioid consumption | 24 hours after surgery
  Dilaudid will be used for analgesia postoperatively. If there is a contraindication to Dilaudid, another opioid will be ordered for analgesia, and doses will subsequently be converted back to Dilaudid equivalent doses for comparison

SECONDARY OUTCOMES:
Cumulative opioid consumption | 4, 8, and 48 hours after surgery
  Dilaudid will be used for analgesia postoperatively. If there is a contraindication to Dilaudid, another opioid will be ordered for analgesia, and doses will subsequently be converted back to Dilaudid equivalent doses for comparison
Verbal pain score (static and dynamic) | PACU, 4, 8, 12, 24, and 48 hours after surgery
  Pain score 0-10 with 10 being worst possible pain
Opioid side effect (nausea/vomiting, pruritus, constipation, urinary retention, sedation) | PACU, 4, 8, 12, 24, and 48 hours after surgery
  Presence of each side effect documented as "yes" or "no". Sedation will be assessed by the Ramsay Sedation Scale.
Overall patient satisfaction | 48 hours after surgery
  Satisfaction rated as: very dissatisfied, dissatisfied, neutral, satisfied, or very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Jacelyn Larson, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Saskatoon City Hospital, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Result] Chelly JE, Ben-David B, Williams BA, Kentor ML. Anesthesia and postoperative analgesia: outcomes following orthopedic surgery. Orthopedics. 2003 Aug;26(8 Suppl):s865-71. doi: 10.3928/0147-7447-20030802-08. PMID 12934742
- [Result] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Result] Birnbaum K, Prescher A, Hessler S, Heller KD. The sensory innervation of the hip joint--an anatomical study. Surg Radiol Anat. 1997;19(6):371-5. doi: 10.1007/BF01628504. PMID 9479711
- [Result] Mitchell ME. Regional anesthesia for hip surgery. Techniques in Regional Anesthesia and Pain Management 3(2): 94-106, 1999.
- [Result] Dalens B, Vanneuville G, Tanguy A. Comparison of the fascia iliaca compartment block with the 3-in-1 block in children. Anesth Analg. 1989 Dec;69(6):705-13. PMID 2589650
- [Result] Dolan J, Williams A, Murney E, Smith M, Kenny GN. Ultrasound guided fascia iliaca block: a comparison with the loss of resistance technique. Reg Anesth Pain Med. 2008 Nov-Dec;33(6):526-31. doi: 10.1016/j.rapm.2008.03.008. PMID 19258967
- [Result] Foss NB, Kristensen BB, Bundgaard M, Bak M, Heiring C, Virkelyst C, Hougaard S, Kehlet H. Fascia iliaca compartment blockade for acute pain control in hip fracture patients: a randomized, placebo-controlled trial. Anesthesiology. 2007 Apr;106(4):773-8. doi: 10.1097/01.anes.0000264764.56544.d2. PMID 17413915
- [Result] Godoy Monzon D, Iserson KV, Vazquez JA. Single fascia iliaca compartment block for post-hip fracture pain relief. J Emerg Med. 2007 Apr;32(3):257-62. doi: 10.1016/j.jemermed.2006.08.011. Epub 2007 Feb 8. PMID 17394987